CLINICAL TRIAL: NCT05421468
Title: Timing of Thyroxine Dose In Ramadan; a Randomized Control Trial
Brief Title: Timing of Thyroxine Dose In Ramadan
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ICT22J-001-01
Record Dates: First submitted 2022-05-27; First posted 2022-06-16 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Hypothyroidism
MeSH Terms: conditions — Hypothyroidism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pre-Iftar (Breaking the fast) (Active Comparator): To take thyroxine at breaking of fast with sip of water then wait 30-60 miuntes to eat iftar (breakfast).
  Interventions: Other: L-Thyroxine time B (5-15 minutes Before dawn)
- Pre-Fajr (Starting the fast) (Experimental): To take thyroxine immediately before start of fast at predawn time regardless of last meal time.
  Interventions: Other: L-Thyroxine time B (5-15 minutes Before dawn)

INTERVENTIONS:
Other: L-Thyroxine time B (5-15 minutes Before dawn) — Taking thyroxine at two different time points in relation to fasting and food intake; just before dawn and start of fast compared to the usual timing of 30-60minutes after the sunset breakfast meal.

SUMMARY:
A Randomized trial comparing two different timing of taking thyroxine in patients with Hypothyroidism during fasting the month of Ramadan.

DETAILED DESCRIPTION:
To date there is debate regarding the best timing of L-thyroxine administration during Ramadan as sufficient evidence is lacking. This study aims to compare two-time points of levothyroxine intake during Ramadan focusing on change in TSH, satisfaction and compliance.

A prospective, randomized, open label, multicenter Study. The first group will be will be instructed to take their L-thyroxin dose as per current guidlines at breaking of fast time (sunset) with sip of water then wait 30-60 minutes to consume Iftar meal. The second group (pre-Fajer prayer), patients are going to be instructed to take L-thyroxin dose immediately before start of fast, i.e. Alfajer (dawn) regardless of Suhoor time. The values of Thyroid stimulating hormone (TSH) will be measured two weeks before Ramadan, and 2-4 weeks after Ramadan for comparison.

ELIGIBILITY:
Inclusion Criteria:

* Saudi patient (males and female) above 18 years with Primary hypothyroidism on levothyroxine replacement who are willing to fast during Ramadan.
* Patients with controlled thyroid function for last 3 months on same dose of levothyroxine.

Exclusion Criteria:

* Pregnant or lactating women.
* Uncontrolled thyroid function test three months prior Ramadan.
* Thyroid cancer patients who require suppressed TSH.
* Central Hypothyroidism, patient with acute illness.
* Patients diagnosed with malabsorption i.e., Celiac Disease, Short bowel, Bariatric surgeries

  * Use of certain Medications like systemic glucocorticoids, activated charcoal, sucralfate, aluminum hydroxide antacid, bile acid sequestrants, iron, calcium carbonate, PPI, rifampicin, and antiepileptic medications
  * Renal or hepatic disease:
  * Creatinine clearance <0.6 ml/s or serum creatinine ≥200 μmol/l
  * Alanine transferase ≥2.5 times the upper limit of normal
  * Active liver disease including jaundice, chronic hepatitis, previous liver transplant
  * Unwillingness to be randomized or to sign informed consent
  * Known Psychiatric Disorders
  * Known uncontrolled substance abuse or alcoholism

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2022-03-14 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Thyroid function | 6 - 8 weeks
  Change in TSH level

CONTACTS AND LOCATIONS:
Locations (2):
- Saudi Arabia (2):
  - Reem Alamoudi, Jeddah
  - KingAbullahIMRC, Jeddah

IPD SHARING:
Plan to Share IPD: Undecided